CLINICAL TRIAL: NCT04076878
Title: Effects of Using the Electrodress Mollii to Reduce Spasticity and Enhance Functioning After Stroke.
Brief Title: Effects of Using the Electrodress Mollii on Spasticity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danderyd Hospital (Other)
Responsible Party: Principal Investigator, Susanne Palmcrantz, Principal Investigator, Danderyd Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mollii for spasticity
Record Dates: First submitted 2019-07-31; First posted 2019-09-03 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Spasticity, Muscle; Stroke; Electric Stimulation Therapy
Keywords: Spasticity; Stroke; Functioning; Disability; Intervention; electrical stimulation therapy
MeSH Terms: conditions — Muscle Spasticity; Stroke

STUDY DESIGN:
Intervention Model Description: Mechanism substudy: explorative single group design with three different stimulation paradigms provided to all participants by double blinded randomisation.
  Clinical substudy: explorative single group design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention in a Mechanism and a Clinical substudy (Experimental): Mechanism substudy: 3 trial sessions ( electrodes set to 1) 20 Hz, 2) 30 Hz, 3) 0 Hz (placebo). Patients and datacollectors were blinded in terms of the randomised order of the treatment at each of the 3 trial sessions ( electrodes set to 1) 20 Hz, 2) 30 Hz, 3) 0 Hz (placebo).
  Clinical substudy: Use of the fitted and individually set body suit, Mollii, in the home setting for 6 weeks
  Interventions: Device: Mollii

INTERVENTIONS:
Device: Mollii — The Mollii method is provided in a tight fitting, whole body suit with multiple electrodes that can be set individually. The Mollii method uses low frequencies and low intensities that evokes sensory input but does not directly elicit muscle contractions. The theoretical background of this treatment method primarily refers to the concept of reciprocal inhibition, i.e. that sensory input from a muscle may inhibit the activation of an antagonistic muscle through the activation of the disynaptic reciprocal Ia inhibitory pathway.

SUMMARY:
Spasticity is a common manifestation of lesions of central motor pathways, such as after stroke, traumatic brain or spinal cord injury and in cerebral palsy and is associated with increased impairments and disabilities. Spasticity may be associated with pain and contractures, caused by muscle weakness, reduced muscle length and volume that add to the disability.Treatments of spasticity comprise physical therapy, pharmacological agents and surgical treatment. Recently, a systematic review concluded that transcutaneous, electric nerve stimulation may have beneficial effects on spasticity and activity performance after stroke, which lends support to the new treatment method Mollii, which will be evaluated in this study.The Mollii suit provides electric stimulation through multiple electrodes places in a tight fitting suit. This study relates to the clinical trials performed at the University department of rehabilitation medicine at Danderyd Hospital in Stockholm and comprises an initial study of effects on spasticity ("Mechanical substudy") and a following, exploratory treatment trial ("Clinical substudy") in patients with spasticity after stroke.

DETAILED DESCRIPTION:
Spasticity is a common manifestation of lesions of central motor pathways, such as after stroke, traumatic brain or spinal cord injury and in cerebral palsy and is associated with increased impairments and disabilities. Spasticity may be associated with pain and contractures, caused by muscle weakness, reduced muscle length and volume that add to the disability.Treatments of spasticity comprise physical therapy, pharmacological agents and surgical treatment. Recently, a systematic review concluded that transcutaneous, electric nerve stimulation may have beneficial effects on spasticity and activity performance after stroke, which lends support to the new treatment method Mollii, which will be evaluated in this study.The Mollii method has been developed by Inervetions, which is a small Swedish med-tech company, and represents an innovative approach for non-invasive electro-stimulation to reduce spasticity and improve motor function. The theoretical background of this treatment method primarily refers to the concept of reciprocal inhibition, i.e. that sensory input from a muscle may inhibit the activation of an antagonistic muscle. Thus, the application of Mollii aims at stimulating a muscle, e.g. the anterior tibial muscle of the lower leg in order to reduce reflex mediated over-activity, i.e. spasticity, in calf muscles by inducing reciprocal inhibition.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants had

* suffered a stroke > 12 months earlier
* were living with hemiplegia affecting the right or the left side of the body including both upper and lower extremity function
* were able to walk with assistance or independently according to the Functional Ambulatory Categories (Holden 1984) with a score of 2-5
* activity in upper extremity was limited according to the Action Research Arm test (ARAT) (Nordin 2014) but could perform a grasp and grip movement
* were > 17 years old, able to understand instructions as well as written and oral study information and could express informed consent

Exclusion Criteria:

* no detected neural component exceeding the cut off for spasticity according to the Neuroflexor (> 3. 4 Newton) in the wrist flexors
* contractures not compatible with performing the Neurofexor test or walking
* any other disorder with an impact on sensorimotor function
* any other severe concomitant disease (such as cancer, cardiovascular, inflammatory or psychiatric disease), uncontrolled epilepsy or blood pressure, major surgery during the last year, any implanted medical devices
* pregnancy
* BMI>35

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Mechanism substudy and Clinical substudy: NeuroFlexor | Mechanism study: To assess change, NeuroFlexor data is recorded before, during and 10 minutes after treatment at each session. Clinical study: To assess change Neuroflexor data is collected before and after the 6 week intervention.
  Measure related to spasticity: The Neuroflexor device comprises a portable computer-controlled step motor system with a lever arm that generates constant velocity movements of the wrist or ankle. The passive resistive force of the wrist or ankle is recorded by a force transducer. The force is then analyzed off-line and the total resistance is separated into mechanical and a neural components using a neuro-biomechanical computerized model. NeuroFlexor neural component reflecting stretch reflex mediated resistance, represents the main outcome. The NeuroFlexor hand (used in mechanism and clinical substudy) and foot module (used in mechansim substudy only) is a valid method that quantifies and distinguishes the genuine spasticity and the mechanical contributions (viscoelastic and soft tissue components) of the resistance opposing a passive stretch.

SECONDARY OUTCOMES:
Mechanism substudy: Surface electromyography | To assess change sEMG are assessed before and after 60 min of treatment at each session.
  Measure related to spasticity: Surface electromyography (sEMG) signal of spastic muscles in the upper and lower limb (flexor carpi radialis, medial gastrocnemius and soleus muscles).
Mechanism substudy: Modified Ashworth scale: | Before and after 60 min of treatment at each session to assess change
  Clinical assessment of spasticity on a 5 point scale ranging from 0= no spasticity to 5= rigidity
Mechanism substudy: Semi structured interview | During the 60 min of treatment at each session
  To assess perceived effects of each intervention
Clinical substudy: the Fugl-Meyer scale | Before and after the 6 week intervention to assess change
  Clinical assessment of motor sensory function of the upper (min 0 p and max 126p) and lower extremity (min 0 p and max 86p). Max point indicates no detected impairment.
Clinical substudy: Modified Ashworth scale | Before and after the 6 week intervention to assess change
  Clinical assessment of spasticity on a 5 point scale ranging from 0= no spasticity to 5= rigidity
Clinical substudy: Barthel Index | Before and after the 6 week intervention to assess change
  Assessment of self-care and mobility (min 0 p and max 100p). Max point indicates independence
Clinical substudy: Berg balance scale | Before and after the 6 week intervention to assess change
  Clinical assessment of balance (max 56p). Max point indicate no limitations in balance.
Clinical substudy: Montreal Cognitive Assessment | Before and after the 6 week intervention to assess change
  Assessment of cognitive function (min 0 p and max 30p). Max point indicate no impairment.
Clinical substudy: Action Research Arm Test | Before and after the 6 week intervention to assess change
  Clinical assessment of activity in upper extremity (max 57 p). Max point indicate no limitation.
Clinical substudy: A digital hand dynamometer | Before and after the 6 week intervention to assess change
  Clinical assessment of grip strength in kilograms.
Clinical substudy: 10 meter walk test | Before and after the 6 week intervention to assess change
  Clinical assessment of walking speed (m/s)
Clinical substudy: 6 min walk test | Before and after the 6 week intervention to assess change
  Clinical assessment of walking endurance (meters)
Clinical substudy: Functional Ambulation Category | Before and after the 6 week intervention to assess change
  Assessment of indedence in walking (min 0 p and max 5p) Max point indicate independence
Clinical substudy: Stroke Impact Scale | Before and after the 6 week intervention to assess change
  Self-perceived functioning and disability (min 0 p and max 100p/item). Max point indicate no perceived disability.
Clinical substudy: Weekly semistructured telephone interview | Weekly during the 6 week intervention
  To assess compliance, perceived effects and adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Palmcrantz, PhD, Principal Investigator — Danderyd Hospital
Locations (1):
- Department of Rehabilitation Medicine, Danderyd Hospital, Danderyd, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gaverth J, Eliasson AC, Kullander K, Borg J, Lindberg PG, Forssberg H. Sensitivity of the NeuroFlexor method to measure change in spasticity after treatment with botulinum toxin A in wrist and finger muscles. J Rehabil Med. 2014 Jul;46(7):629-34. doi: 10.2340/16501977-1824. PMID 24850135
- [Background] Gaverth J, Sandgren M, Lindberg PG, Forssberg H, Eliasson AC. Test-retest and inter-rater reliability of a method to measure wrist and finger spasticity. J Rehabil Med. 2013 Jul;45(7):630-6. doi: 10.2340/16501977-1160. PMID 23695917
- [Background] Lindberg PG, Gaverth J, Islam M, Fagergren A, Borg J, Forssberg H. Validation of a new biomechanical model to measure muscle tone in spastic muscles. Neurorehabil Neural Repair. 2011 Sep;25(7):617-25. doi: 10.1177/1545968311403494. Epub 2011 Apr 13. PMID 21490269
- [Derived] Pennati GV, Bergling H, Carment L, Borg J, Lindberg PG, Palmcrantz S. Effects of 60 Min Electrostimulation With the EXOPULSE Mollii Suit on Objective Signs of Spasticity. Front Neurol. 2021 Oct 15;12:706610. doi: 10.3389/fneur.2021.706610. eCollection 2021. PMID 34721255
- [Derived] Palmcrantz S, Pennati GV, Bergling H, Borg J. Feasibility and potential effects of using the electro-dress Mollii on spasticity and functioning in chronic stroke. J Neuroeng Rehabil. 2020 Aug 10;17(1):109. doi: 10.1186/s12984-020-00740-z. PMID 32778118